CLINICAL TRIAL: NCT06453902
Title: A Single-arm, Open-label, Multi-center Phase II Study Evaluating Efficacy and Safety of TGRX-678 in CML-AP Patients Relapsed or Refractory From 3rd-generation TKI Treatment
Brief Title: TGRX-678 Chinese Phase II in Chronic Myelogenous Leukemia (CML) Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen TargetRx, Inc. (Industry)
Collaborators: Peking University People's Hospital (Other); Henan Cancer Hospital (Other Government); Nanfang Hospital, Southern Medical University (Other); The First Affiliated Hospital of Soochow University (Other); Chinese Academy of Medical Sciences (Other); First Affiliated Hospital of Zhejiang University (Other); Shenzhen Second People's Hospital (Other); Ruijin Hospital (Other); Shengjing Hospital (Other); Tongji Medical College,Huazhong University of Science &Techonlogy (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGRX-678-2001
Record Dates: First submitted 2024-05-28; First posted 2024-06-12 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Chronic Myeloid Leukemia; Accelerated Phase CML
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Accelerated Phase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: TGRX-678 (Experimental): All patients with CML-AP to be treated with TGRX-678. Patients with T315I mutation or without T315I mutation will be assigned into separate cohorts for evaluation
  Interventions: Drug: TGRX-678

INTERVENTIONS:
Drug: TGRX-678 — All patients will be given TGRX-678 240 mg once daily. TGRX-678 is to be taken orally

SUMMARY:
A Phase II study evaluating the safety and efficacy of TGRX-678 in Chronic Myelogenous Leukemia (CML) patients in Accelerated phase (AP) and are relapsed or refractory from third-generation Tyrosine Kinase Inhibitor (TKI) treatment

DETAILED DESCRIPTION:
This Phase II study is of single-arm, open-label and multi-center designs to study safety and efficacy profiles of TGRX-678 in CML-AP patients. Patients need to have medical history of failing treatment(s) from third-generation TKI drugs. Patients with or without T315I mutation is enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Willing to consent
* 18 years of age or above at time of screening; both sexes eligible
* Relapsed or refactory from 3rd-generation Tyrosine kinase inhibitor (TKI) treatment
* For patients without T315I mutation, the patients must received 1st, 2nd and 3rd generation TKI
* For patients with T315I mutation, the patients much received Olverembatinib or Ponatinib treatment
* Diagnosis of CML-AP by bone marrow morphological test, molecular biology test or cytogenetic tests
* ECOG score </=2
* Minimum life expectancy of at least 3 months
* Adequate hematological indicators
* Adequate kidney function
* Adequate liver function
* Adequate coagulation function
* Adequate pancreatic function
* Adequate QTc interval as confirmed by electrocardiogram (ECG) test
* Negative pregnancy result at screening for female patients of child-bearing potential
* Willing to take contraceptive measure during the study (For male and female patients of child-bearing potential)

Exclusion Criteria:

* Reception of TKI treatment or presence of unrecovered TKI treatment related non-hematological adverse events within 7 days of first dose
* Reception of other anti-tumor treatments
* In need for immune suppressive treatment
* Usage of drugs associated with Torsades de Pointes within 1 months before screening
* Presence of other medical conditions that require using treatment that may have drug-drug interaction with the investigational drug
* History of hemapoietic stem cell transplant
* Presence of active central nervous system conditions
* CML-AP patients who already reached major hematological response
* CML-AP patients who used to progress to Blast Phase (BP)
* Presence or having uncontrolled condition for cardiovascular diseases
* History of any heart or cardiovascular conditions (except for patients with hypertension which is controlled by anti-hypertensive drugs, and blood pressure is controlled at no higher than 160/100 mmHg for 1 months before screening)
* Usage of any Traditional Chinese Medicine indicated for anti-tumor purpose 2 weeks before first dose
* Severe hemorrhagic disease unrelated to CML
* History of severe cardiovascular condition during past TKI treatment for CML
* History of pancreatic inflammation or alcohol abuse within 3 years before first dose
* Uncontrolled Hypertriglyceridemia
* Presence of malabsorption or other conditions that may affect drug absorption
* Diagnosis of other primary malignant tumor within 5 years
* Reception of major surgery 14 days before first dose
* Presence of continuous or active infection (including HIV, hepatitis B, hepatitis C)
* Presence of other conditions that the investigators or medical monitor deem unfit for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Major Hematologic Response (MaHR) | At screening, on Day 1 of every treatment cycle (each cycle is 28 days) and at end of treatment; average of study duration is 3.5 years
  Number of patients who reached, and rate of occurence of major hematologic response, including those who reached complete hematologic response (CHR) or no evidence of leukemia (NEL). CHR and NEL are defined per China national treatment guideline for CML (ver. 2022). Indicators for hematologic responses will be obtained via peripheral blood tests.

SECONDARY OUTCOMES:
Cytogenetic Response | At screening, on Day 1 of cycle 2, cycle 4 and every 3 cycles afterwards of the treatment cycle (each cycle is 28 days) and at the end of treatment; average of study duration is 3.5 years
  Number of patients who reached, and rate of occurence of cytogenetic response, including those with major cytogenetic response (MCyR) or complete cytogenetic response (CCyR). Cytogenetic responses are defined per China national treatment guideline for CML (ver. 2022). Indicators for cytogenetic responses will be obtained via bone marrow biopsy.
Major Molecular Response (MMR) | At screening, on Day 1 of cycle 2, cycle 4 and every 3 cycles afterwards of the treatment cycle (each cycle is 28 days) and at the end of treatment; average of study duration is 3.5 years
  Number of patients who reached, and rate of occurence of MMR. Cytogenetic response is defined per China national treatment guideline for CML (ver. 2022). Indicators for molecular responses will be obtained via genetic testing on transcript levels of BCR-ABL gene.
Time to Response (TTR) | At screening, on Day 1 of cycle 2, cycle 4 and every 3 cycles afterwards of the treatment cycle (each cycle is 28 days) and at the end of treatment; average of study duration is 3.5 years
  TTR defined by the time from the start of treatment to the first efficacy response; TTR as evaluated by investigator
Duration of Response (DOR) | At screening, on Day 1 of cycle 2, cycle 4 and every 3 cycles afterwards of the treatment cycle (each cycle is 28 days) and at the end of treatment; average of study duration is 3.5 years
  DOR defined as the duration from first occurence of treatment response to progressive disease/relapse; DOR as evaluated by investigator
Progression Free Survival (PFS) | At screening, on Day 1 of cycle 2, cycle 4 and every 3 cycles afterwards of the treatment cycle (each cycle is 28 days) and at the end of treatment; average of study duration is 3.5 years
  PFS defined as the time from enrollment to progressive disease or death of any cause; PFS as evaluated by investigator.
Overall Survival (OS) | At screening, on Day 1 of cycle 2, cycle 4 and every 3 cycles afterwards of the treatment cycle (each cycle is 28 days) and at the end of treatment; average of study duration is 3.5 years
  OS defined as the time from enrollment to death of any cause; OS as evaluated by investigator
Treatment Emergent Adverse Event (TEAE) | Through completion of the study, an average of 3.5 years
  To record and analyse the occurence and frequency of adverse events during the study

CONTACTS AND LOCATIONS:
Overall Officials: Qian Jiang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China